CLINICAL TRIAL: NCT01041391
Title: Lumbar Disc Herniation Outcome Measures-Surgical Versus Non-Operative Treatment
Brief Title: Lumbar Disc Herniation Outcome Measures
Status: Terminated | Type: Observational
Why Stopped: Slow/low enrollment
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Principal Investigator, William Lavelle, Associate Professor, State University of New York - Upstate Medical University
Other Study IDs: 5812-LSS
Record Dates: First submitted 2009-11-18; First posted 2009-12-31 (Estimated); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Lumbar Intervertebral Disc Herniation
Keywords: Surgical intervention vs Non-Surgical intervention
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Surgical treatment for Lumbar disc herniation: Patients who had or will have surgery for Lumbar disc herniation
  Interventions: Procedure: Discectomy-lumbar spine
- Non-surgical treatment for Lumbar disc herniation: Patients that have chosen conservative treatment for lumbar disc herniation

INTERVENTIONS:
Procedure: Discectomy-lumbar spine — Lumbar intervertebral discectomy performed on patients with herniated disc that chose to have surgical intervention
  Groups: Surgical treatment for Lumbar disc herniation

SUMMARY:
This study is being conducted to examine outcome measurements on patients who undergo surgery to removed a damage lumbar spine disc versus those that chose not to have surgery. These outcomes are based on patient responses to quality of life and pain questionnaires.

DETAILED DESCRIPTION:
Lumbar discectomy is the most common surgical procedure performed for back and leg symptoms in US patients, but the efficacy of the procedure relative to non-operative care remains controversial.

Several studies have compared surgical and non-operative treatment of patients with herniated discs, but baseline differences between treatment groups, small sample sizes, or lack of validated outcome measures in these studies limit evident-based conclusions regarding optimal treatment.

There is increasing emphasis on the use of health-related quality of life(QOL)outcome measures to determine the efficacy of treatment, particularly for diseases that are not life threatening but affect the patient's QOL. In the treatment of lumbar disc herniation, the Medical Outcomes Study Short Form (SF-36), Oswestry Disability Index (ODI) and Visual Analog Scale (VAS), are validated and common scales that are used to measure treatment outcomes.

Information is routinely collected on activity limitations in the course of the doctor's assessment of the patient, however, the data may not always be collected in a standardized format that yields measurement with known reliability and validity. Standardized self-report questionnaires provide a convenient method of collecting and synthesizing a large amount of information on the pain, activity limitation and general health status of each patient.

The objective of this prospective study is to evaluate the efficacy of surgery for lumbar intervertebral disc herniations using the SF-36, ODI and VAS as primary outcome measures. Patients experiencing acute or chronic lumbar spine pain in the Orthopedic practice will be given a choice to participate in this study. On patient's who wish to participate, the data will be collected and entered into the REMARK OMR 7 database, and evaluated for outcomes.

This study is for current patients in the Upstate Orthopedic office.

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 18 years of age and no older than 90 years of age
* Must have diagnosis of Lumbar disc herniation
* Must be able to understand English, and willing to consent to data collection
* Must be a current patient in our practice

Exclusion Criteria:

* Prisoner
* Unable to complete questionnaires

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in the SUNY Upstate Orthopedic Surgery department
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2009-05; Primary Completion 2013-01-13 (Actual); Study Completion 2013-01-13 (Actual)

PRIMARY OUTCOMES:
The efficacy of surgery for lumbar intervertebral disc herniation vs non-operative treatment, using self-report questionnaires Short form 36, Visual Analog Scale and Oswestry Disability Index at baseline (prior to surgery) and all subsequent visits | baseline (prior to surgery) & 12 mos post op.
  data will be collected at each office visit, regardless of time point

CONTACTS AND LOCATIONS:
Overall Officials: William F. Lavelle, MD, Principal Investigator — State University of New York - Upstate Medical University
Locations (1):
- SUNY Upstate Medical University-Department of Orthopedics, Syracuse, New York, United States